CLINICAL TRIAL: NCT01807247
Title: Evaluation of the Short Effects of a Rehabilitation Session on Gait Parameters in Patients With a Lesion of the Central Nervous System
Brief Title: Short Effects of a Rehabilitation Session on Gait in Patients With CNS
Status: Completed | Type: Observational
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Principal Investigator, Nicolas ROCHE, MDPHD, Centre d'Investigation Clinique et Technologique 805
Other Study IDs: 2011-A01487-34
Record Dates: First submitted 2013-03-07; First posted 2013-03-08 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2013-03

CONDITIONS: Spastic Gait; Fall Due to Failure of Support; Fatigue
Keywords: Strengthening muscle; Central nervous system diseases; Gait
MeSH Terms: conditions — Gait Disorders, Neurologic; Fatigue; Central Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Hemiparetic: Intensive lower limbs muscles strengthening
  Interventions: Procedure: Intensive lower limbs muscles strengthening
- Spinal cord injury: Intensive lower limbs muscles strengthening
  Interventions: Procedure: Intensive lower limbs muscles strengthening
- Multiple sclerosis: Intensive lower limbs muscles strengthening
  Interventions: Procedure: Intensive lower limbs muscles strengthening

INTERVENTIONS:
Procedure: Intensive lower limbs muscles strengthening

SUMMARY:
The aim of the study is to evaluate the short effects of a two rehabilitation session commonly performed in physical therapy,

1. muscle strengthening of the lower limbs and
2. effort reconditioning with cyclo ergometer, on gait characteristics (kinematics, kinetics and electromyographic) in patients with central nervous system lesion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged ≥ 18 years receiving a motor rehabilitation in the service
* Hemiplegia after stroke or paraplegia incomplete ASIA C or D or multiple sclerosis (EPSS <5).
* Walking with or without technical assistance
* Patients who received and signed information and informed consent
* Patient who received physiotherapy session for rehabilitation of the lower limbs
* Patients able to perform the entire study

Exclusion Criteria:

* Patient with safety measure
* Pregnant women, breastfeeding
* Patient who has received botulinum toxin injection of in the lower limbs between 3 weeks and 2 months prior to inclusion in the study
* Bilateral Brain damage, cerebellar syndrome, apraxia, severe aphasia
* Orthopedic complications preventing walking
* Patients who participated in a clinical study within 3 months prior to inclusion • No affiliation to a social security scheme (beneficiary or assignee)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population includes patients with various lesions of central nervous system such as post-stroke patients with hemiparesis, patients with spinal cord injury and patients with mutiple sclerosis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of functional capacity after rehabilitation session using functional tests such as 6 minutes walking test and timed up and go | 30 min
  clinical exam, timed up and go, stair test, 6 minutes walking test

SECONDARY OUTCOMES:
Evaluation of gait pattern and muscle activation patterns during video and EMG analyzes. | 1 hour
  EMG analysis of rectus femoris, hamstrings, tibialis anterior and soleus

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas ROCHE, MDPHD, Principal Investigator — Hôpital RAYMOND POINCARE
Locations (1):
- Hopital Raymond Poincare, Garches, Garches, France